CLINICAL TRIAL: NCT05259683
Title: Validating Clinical Decision Aids for the Assessment and Management of Febrile Infants Presenting to Emergency Care in the UK and Ireland.
Brief Title: Febrile Infant Diagnostic Assessment and Outcome Study
Acronym: FIDO
Status: Completed | Type: Observational
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Thomas Waterfield, Clinical Lecturer, Queen's University, Belfast
Other Study IDs: 278080
Record Dates: First submitted 2022-02-10; First posted 2022-02-28 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Urinary Tract Infections; Meningitis; Sepsis; Bacterial Infections
MeSH Terms: conditions — Urinary Tract Infections; Meningitis; Sepsis; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1ml of residual blood plasma collected during routine phlebotomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Febrile infants under 3 months of age represent a high risk group for invasive bacterial infection (IBI) and UTI with approximately 10-20% having bacteremia, meningitis or urinary tract infection. The assessment of febrile infants is challenging, and current National Institute for Health and Care Excellence (NICE) guidance advocates a cautious approach with the majority of infants requiring a septic screen, parenteral broad-spectrum antibiotics, and admission to hospital. Internationally there is significant variation in the approach to febrile infants with European and USA guidance advocating a tailored approach based on clinical features and biomarker testing. None of the available clinical decision aids (CDA) have been validated in a UK and Irish cohort. The main objectives of the FIDO study are to report performance accuracy of CDA in a UK (United Kingdom) and Irish population, and describe the aetiology of SBI in young infants.

The FIDO study is a prospective observational cohort study of infants under 90 days of age with a measured fever greater than 38 Centrigrade within 24 hours of presentation. The study will run for approximately 12 months and recruit a minimum of 1000 participants.Symptoms, clinical features and laboratory results will be recorded on an electronic case report form (CRF) by the attending clinician.

DETAILED DESCRIPTION:
Background

Infants below three months of age are at high risk of invasive bacterial infections (IBI) and urinary tract infections (UTI). Recent studies have reported the combined rate of IBI and UTI in the range of 10 - 20% , with IBI (bacteremia and meningitis) account for to up to 3% of the total. Unlike older children infants regularly appear well or have non-specific features despite having an IBI or UTI, with history and physical examination alone not sufficient to detect all cases. Furthermore, the clinical differentiation between fever caused by bacteria and viruses is most challenging in the less than three month age group. The majority of children still have self-limiting illness in this age group making risk assessment challenging for clinicians.

The ideal approach to the assessment and management of febrile infants is not clear, as exemplified by the contrasting approaches advocated by the National Institute for Health and Care Excellence (NICE). The NICE guideline 51 (NG51) "Sepsis: recognition, diagnosis and early management" advises that all febrile infants (under 3 months of age) receive parenteral antibiotics immediately whereas NICE guideline 143 (NG143) "Fever in under 5s: assessment and initial management" suggests a tailored approach based on clinical assessment and laboratory testing. The recently proposed British Society for Antimicrobial Chemotherapy (BSAC) guidance also supports a tailored approach similar to the NICE guideline NG143. The primary aim of this study is to prospectively validate these CDA.

Objectives Primary Objectives

* Report the aetiology of IBI in febrile infants under three months in the UK and Ireland.
* Describe the clinical and laboratory predictors of IBI in febrile infants under three months of age.
* Report the performance of tailored CDAs to correctly identify a cohort suitable for management without parenteral antibiotics.
* Report the performance of tailored CDAs to correctly identify a cohort suitable for management without lumbar puncture.

Secondary Objectives

* Report a cost analysis for different CDAs.
* Report parents/guardians' and clinicians' views on how best to communicate different treatment strategies, including the risks and benefits of each.

Study Design A multicentre observational prospective cohort study in the UK and Ireland conducted via Paediatric Emergency Research in the UK and Ireland (PERUKI).

Study Population All infants 90 days of age and under with a fever of greater than 38 Centigrade during their time in the Emergency Department (ED) or Assessment Unit (AU) or with a history of fever of greater than 38 Centigrade recorded by anyone via any thermometer type within the last 24 hours. There are no exclusion criteria, but data will be recorded regarding gestational age, antenatal complications, underlying health conditions and recent admissions to hospital.

Setting PERUKI sites across the UK and Ireland.

Screening Eligible participants will be screened by appropriately trained clinical staff, using the case report form (CRF). The CRF will be used to record anonymised non-personal data such as baseline demographic data, clinical features and initial examination findings.

Procedures All eligible participants will be enrolled. In all instances routine care will not be interrupted. Where possible an additional 1ml of blood will be taken and stored for PCT testing. This blood will be collected during routine phlebotomy. There will be no additional phlebotomy events beyond those required for routine clinical care. Seven days after discharge the CRF will be completed by a trained member of the local study team. This will involve reviewing the medical records and a phone call (maximum of three attempts) to the parent/guardian to determine if there had been any subsequent unplanned re-attendances to hospital.

Reference Standards The reference standard is the diagnosis of IBI (meningitis/bacteremia) and urinary tract infection (excluding contaminants).

Urinary Tract Infection (UTI) will be confirmed by >100,000 CFU/ml of a single organism from a single clean urine (clean catch, suprapubic aspiration, urethral catheter specimen) or >100,000 Colony Forming Units (CFU)/ml of the same single organism from two non-clean urines (pads, bags, cotton wool) and the presence of pyuria (>5 white blood cells per high powered-field) on laboratory microscopy.

Meningitis will be confirmed by culture or molecular testing of cerebrospinal fluid (CSF). The reference standard test will be performed by staff blinded to the clinical data and suspected diagnosis.

Bacteremia will be confirmed by culture or molecular testing of blood. The reference standard test will be performed by staff blinded to the clinical data and suspected diagnosis.

Contaminants include coagulase negative Staphylococcus, Propionibacterium acnes, Streptococcus viridans, or Diphtheroides. A list of all suspected contaminants will be provided at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* All infants 90 days of age and under with a fever of greater than 38 Centigrade during their time in the Emergency Department (ED) or Assessment Unit (AU) or with a history of fever of greater than 38 Centigrade recorded by anyone via any thermometer type within the last 24 hours.

Exclusion Criteria:

* None

Max Age: 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants attending paediatric emergency care in the United Kingdom and Ireland
Sampling Method: Non-Probability Sample
Enrollment: 2076 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Urinary Tract Infection | 7 days of attendance
  Urinary Tract Infection (UTI) will be confirmed by >100,000 CFU/ml of a single organism from a single clean urine (clean catch, suprapubic aspiration, urethral catheter specimen) or >100,000 CFU/ml of the same single organism from two non-clean urine samples (pads, bags, cotton wool) and pyuria (>5 white blood cells per high-powered field) on laboratory microscopy.
Bacterial Meningitis | 7 days of attendance
  Meningitis will be confirmed by culture or molecular testing of cerebrospinal fluid (CSF).The reference standard test will be performed by staff blinded to the clinical data and suspected diagnosis.
Bacteriaemia | 7 days of attendance
  Bacteremia will be confirmed by bacterial culture or molecular testing of blood using quantitative polymerase chain reaction. The reference standard test will be performed by staff blinded to the clinical data and suspected diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Waterfield, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Queen's University Belfast, Belfast, Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
To be determined

REFERENCES:
- [Derived] Umana E, Mills C, Norman-Bruce H, Mitchell H, McFetridge L, Lynn F, McKeeman G, Foster S, Barrett MJ, Roland D, Lyttle MD, Watson C, Waterfield T; Paediatric Emergency Research in the UK and Ireland (PERUKI). Performance of clinical decision aids (CDA) for the care of young febrile infants: a multicentre prospective cohort study conducted in the UK and Ireland. EClinicalMedicine. 2024 Nov 27;78:102961. doi: 10.1016/j.eclinm.2024.102961. eCollection 2024 Dec. PMID 39677360
- [Derived] Evans J, Umana E, Waterfield T; FIDO Study Group in collaboration with PERUKI. Respiratory viral testing for young febrile infants presenting to emergency care: a planned secondary analysis of the Febrile Infants Diagnostic assessment and Outcome (FIDO) prospective observational cohort study. Arch Dis Child. 2024 Nov 19;109(12):988-993. doi: 10.1136/archdischild-2024-327567. PMID 39357988
- [Derived] Wilson K, Umana E, McCleary D, Waterfield T, Woolfall K. Exploring communication preferences and risk thresholds of clinicians and parents of febrile infants under 90 days presenting to the emergency department: a qualitative study. Arch Dis Child. 2024 Oct 18;109(11):886-893. doi: 10.1136/archdischild-2023-326727. PMID 38986575
- [Derived] Umana E, Mills C, Norman-Bruce H, Wilson K, Mitchell H, McFetridge L, Woolfall K, Lynn FA, McKeeman G, Foster S, Barrett M, Roland D, Lyttle MD, Watson C, Waterfield T. Applying clinical decision aids for the assessment and management of febrile infants presenting to emergency care in the UK and Ireland: Febrile Infant Diagnostic Assessment and Outcome (FIDO) Study protocol. BMJ Open. 2023 Sep 20;13(9):e075823. doi: 10.1136/bmjopen-2023-075823. PMID 37730397